CLINICAL TRIAL: NCT07251192
Title: Testing the Efficacy of a New Intervention for High Intensity Drinking Among Emerging Adults
Brief Title: Social Media Intervention for Risky Drinking
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Erin Bonar, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HUM00285001; R01AA032680 (NIH)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Drinking Behavior
MeSH Terms: conditions — Drinking Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Link to an educational website about alcohol; link to resources.
- Social media messaging (Experimental): Health coaching via social media for 8 weeks
  Interventions: Behavioral: Social media messaging

INTERVENTIONS:
Behavioral: Social media messaging — A motivational interviewing-based intervention delivered via private health coaching on social media for 8 weeks
  Arms: Social media messaging

SUMMARY:
This study is being completed to test prevention methods to promote wellness and reduce risky behaviors, including the use of substances such as alcohol and other drugs. This study will help the study team learn about ways of delivering this information that is both appealing and helpful to young adults.

ELIGIBILITY:
Inclusion Criteria:

Reside in the United States of America (USA) Be able to read English, view, and click on a social media advertisement. Self-reported past-month high-intensity drinking (HID) Regular Snapchat use (at least 3 days/week).

Exclusion Criteria:

Fail identity verification (e.g., IP address, survey completion time) Do not provide sufficient contact information Participated in prior pilot study of same intervention

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Typical weekly drinking (Daily Drinking Questionnaire) | 4-, 8-, and 12-months
  Change in total typical weekly drinks from baseline to follow-up

SECONDARY OUTCOMES:
Alcohol Use Severity (AUDIT-C) | 4-, 8-, and 12-months
  Change in AUDIT-C score from baseline to follow-up
Depression symptoms (PHQ-8) | 4-, 8-, and 12-months
  Change in depression symptom severity as measured by PHQ-8
Anxiety Symptoms (GAD-7) | 4-, 8-, and 12-months
  Change in anxiety symptom severity as measured by GAD-7

CONTACTS AND LOCATIONS:
Overall Officials: Erin E Bonar, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
With participant consent, de-identified data are shared with a data repository with restricted access for future research, as required by the NIAAA.
Supporting Information: Study Protocol, SAP